CLINICAL TRIAL: NCT01180530
Title: A Multicentre, Observational Study of NovoPen Echo® on Safety and Treatment Satisfaction of Insulin Therapy in Children and Adolescents With Diabetes Mellitus
Brief Title: Observational Study of NovoPen Echo® on Safety and Treatment Satisfaction in Children and Adolescents With Type 1 Diabetes
Acronym: REMIND™
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: PDS328-3741; U1111-1113-5037 (Other: WHO)
Record Dates: First submitted 2010-08-06; First posted 2010-08-12 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Delivery Systems
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Device: NovoPen Echo®

INTERVENTIONS:
Device: NovoPen Echo® — Prescribed insulin treatment delivered by NovoPen Echo®

SUMMARY:
This study is conducted in Asia, Europe and North America. The aim of this observational study is to evaluate the safety of NovoPen Echo® by collecting safety information (incidence of technical complaints related to adverse reactions). Study duration: 12-18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children/adolescents with type 1 diabetes mellitus
* After the participating physician's decision has been made to initiate treatment with NovoPen Echo®, any patient who meets all the inclusion criteria and does not meet any of the exclusion criteria, is eligible to participate
* Use of insulin pen or syringes for at least 12 months

Exclusion Criteria:

* Insulin pump or Insuflon® users
* Any disease or condition in children/adolescents which might interfere with the study at the individual physician's discretion

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Any child or adolescent with type 1 diabetes who has just started using NovoPen Echo® is eligible. The selection of the patients will be at discretion of the individual physician.
Sampling Method: Non-Probability Sample
Enrollment: 358 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The incidence of technical complaints related to adverse reactions | after 12-18 weeks (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (4):
- Novo Nordisk Investigational Site, Mississauga, Canada
- Novo Nordisk Investigational Site, Espoo, Finland
- Novo Nordisk Investigational Site, Kfar Saba, Israel
- Novo Nordisk Investigational Site, Malmo, Sweden

REFERENCES:
- [Result] Hansen B, Lilleore SK, Ter-Borch G. Needle with a novel attachment versus conventional screw-thread needles: a preference and usability test among adults with diabetes and impaired manual dexterity. Diabetes Technol Ther. 2011 May;13(5):579-85. doi: 10.1089/dia.2010.0214. Epub 2011 Mar 15. PMID 21406015
- [Result] Adolfsson P, Veijola R, Huot C, Hansen HD, Lademann JB, Phillip M. Safety and patient perception of an insulin pen with simple memory function for children and adolescents with type 1 diabetes--the REMIND study. Curr Med Res Opin. 2012 Sep;28(9):1455-63. doi: 10.1185/03007995.2012.698258. Epub 2012 Jul 27. PMID 22640459
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com